CLINICAL TRIAL: NCT06317272
Title: BReath hOld TecHniquEs for Radiotherapy of Esophageal Carcinoma; a Feasibility Study - Part 1
Brief Title: BReath Hold TecHniquEs for Radiotherapy of Esophageal Carcinoma
Acronym: BROTHER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor inclusion
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RT2016-04-BROTHER Part 1
Record Dates: First submitted 2024-02-27; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: The participating patients will undergo weekly (during radiotherapy treatment) 2 CTs in DIBH; one using ABC and one using voluntary coaching (VC).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABC DIBH (Active Comparator): Active Breathing Controlled (ABC) technique for deep breath inspiration hold (DIBH)
  Interventions: Other: DIBH using ABC technique
- VC DIBH (Experimental): Voluntary Coached (VC) technique for deep breath inspiration hold (DIBH)
  Interventions: Other: DIBH using VC technique

INTERVENTIONS:
Other: DIBH using ABC technique — Deep breath inspiration hold (DIBH) using Active Breathing Control (ABC) technique
  Arms: ABC DIBH
Other: DIBH using VC technique — Deep breath inspiration hold (DIBH) using Voluntary Coaching (VC) technique
  Arms: VC DIBH

SUMMARY:
The main objective of the first part of the study is to determine the most optimal method for DIBH (active breathing control vs voluntary coached) and its reproducibility. Based on these findings, one of these methods will be selected for part 2 of this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven esophageal cancer of the mid or distal esophagus
* Scheduled for external-beam photon radiotherapy with curative intention.
* WHO 0-2.
* Age >= 18 years
* Written informed consent.

Exclusion Criteria:

* Serious respiratory distress
* Contra-indication for fiducial marker placement
* Noncompliance with any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Feasibility DIBH | Week 1, 2, 3, 4, 5 during radiotherapy
  Breath hold maintained for >20 seconds
Reproducibility DIBH | Week 1, 2, 3, 4, 5 during radiotherapy
  Diaphragm dome position within 1cm of the baseline CT Target coverage >94% of the prescribed dose (at 98% of the ITV)

CONTACTS AND LOCATIONS:
Overall Officials: C.T. Muijs, MD, PhD, Principal Investigator — UMC Groningen
Locations (1):
- UMC Groningen, Groningen, Netherlands